CLINICAL TRIAL: NCT07272954
Title: Effects of Ultrasound-Guided Stellate Ganglion Block and Transcutaneous Auricular Vagus Nerve Stimulation on Sleep Quality After Radical Mastectomy for Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Principal Investigator, Qing-he Zhou, PHD, Affiliated Hospital of Jiaxing University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025-LP-777
Record Dates: First submitted 2025-11-22; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Sleep Disorder (Disorder)
Keywords: taVNS
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate Ganglion Block（SGB） (Active Comparator): Before the induction of anesthesia in the operating room, a skilled anesthesiologist performed a SGB under sterile conditions using real-time ultrasound in a blind grouping manner.
  Interventions: Procedure: SGB
- transcutaneous vagus nerve stimulation（taVNS） (Experimental): Three stimulations of transcutaneous auricular vagus nerve stimulation (taVNS) were administered to the patients
  Interventions: Device: taVNS

INTERVENTIONS:
Procedure: SGB — Before the induction of anesthesia in the operating room, a skilled anesthesiologist performed a SGB under sterile conditions using real-time ultrasound in a blind grouping manner. The patient was positioned supine with the neck slightly rotated to the left. A linear probe (6-13 MHz) was placed on the neck to clearly visualize the carotid artery, internal jugular vein, vertebral artery, vagus nerve, thyroid gland, esophagus, scalene muscles, and the anterior scalene muscle at the C6 level. Subsequently, a 48mm, 20-gauge needle was inserted in a "plane" direction into the prevertebral fascia of the anterior scalene muscle. After the needle tip penetrated the prevertebral fascia and negative pressure aspiration was confirmed, 3ml of 0.5% ropivacaine was injected, and the diffusion of the local anesthetic was observed under ultrasound guidance.
  Arms: Stellate Ganglion Block（SGB）
Device: taVNS — Three stimulations of transcutaneous auricular vagus nerve stimulation (taVNS) were administered to the patients: ① According to the manufacturer's recommendations and previous studies [32], the initial adjustment required electrical stimulation to penetrate the skin barrier. The first intervention was conducted one day prior to the surgery, with an initial electrical stimulation frequency set at 30 Hz and a pulse width of 300 μs. The frequency and pulse width were adjusted based on the individual patient's sensations until the maximum tolerable current stimulation was reached without discomfort, lasting for 30 minutes; ② The second intervention occurred immediately after the patient was connected to the monitoring equipment in the operating room, once their vital signs were confirmed to be within normal ranges. The same stimulation frequency as the first intervention was applied for 30 minutes; ③ The third intervention was administered in the recovery room after the patient's surgery
  Arms: transcutaneous vagus nerve stimulation（taVNS）

SUMMARY:
This study aims to design a prospective, randomized, controlled, dual-center, non-inferiority trial to compare the effects of ultrasound-guided sympathetic ganglion block (SGB) and transcutaneous auricular vagus nerve stimulation (taVNS) on sleep quality following radical mastectomy for breast cancer. The objective is to explore whether non-invasive neuromodulation for sleep is non-inferior to invasive neuromodulation. Participants will be randomly assigned to receive either SGB or taVNS treatment. Sleep quality will be assessed using an actigraphy device and sleep scales within four days post-surgery, and the incidence of sleep disturbances will be followed up within 30 days post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-80 years who underwent radical surgery for breast cancer
* ASA I-III

Exclusion Criteria:

* 1. Patients with coagulation dysfunction;
* Patients with suspected regional infection leading to severe nerve damage in the affected limb;
* Patients with congenital heart disease, coronary artery disease, myocardial infarction, severe cardiac conduction block, or those with implanted cardiac pacemakers;
* Patients with severe neurological disorders such as cerebral infarction, cerebral hemorrhage, or stroke;
* Patients with pain, lesions, infections, or unresolved external ear trauma in the area near the external ear;
* Patients with severe mental illness or a history of substance abuse related to analgesics or psychiatric medications;
* Patients with allergies to local anesthetics such as lidocaine or ropivacaine, as well as to general anesthetics;
* Patients and their families who refuse surgical anesthesia and those unable to complete the survey questionnaire.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 136 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Total Sleep Time on the First Night Post-Surgery | the First Night Post-Surgery
  Total Sleep Time Monitored by Actigraphy on the First Night Post-Surgery

SECONDARY OUTCOMES:
Total sleep time from the second to the fourth night post-surgery | the second to the fourth night post-surgery
  Total sleep time each night from the second to the fourth night post-surgery by Actigraphy
Assessment of sleep quality during the first four nights postoperatively | during the first four nights postoperatively
  Assessment of sleep quality using the Richards-Campbell Sleep Questionnaire(RCSQ) sleep questionnaire during the first four nights postoperatively. The total score is 150 points, with the minimum score being 0 points. A higher score indicates better postoperative sleep quality.
sleep quality and the incidence of sleep disturbances on the 30th postoperative day | On the 30th postoperative day
  On the 30th postoperative day, the Pittsburgh Sleep Quality Index (PSQI) will be used to assess subjective sleep quality and the incidence of sleep disturbances.The score ranges from 0 to 21 points, with higher scores indicating worse postoperative sleep quality.A score greater than 7 indicates the presence of sleep disturbance.
The incidence of all complications and mortality within 72 hours postoperatively | within 72 hours postoperatively
  The incidence of all complications and mortality within 72 hours postoperatively
Quality of Recovery score at 24 hours postoperatively (QoR-15). | at 24 hours postoperatively
  Quality of Recovery score at 24 hours postoperatively (QoR-15). The score ranges from 0 to 150 points, with higher scores indicating better postoperative recovery quality.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol